CLINICAL TRIAL: NCT01523158
Title: An Open Study to Investigate the Effects of Injection Immunotherapy on Allergen-specific T and B Cell Responses in Adult Patients With Seasonal Allergic Rhinitis.
Brief Title: Mechanisms of Allergen Immunotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: R and D approval not forthcoming
Sponsor: Royal Sussex County Hospital (Other)
Responsible Party: Principal Investigator, Nicola Gray, Clinical Research Fellow, Royal Sussex County Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12/014/TAR
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunotherapy (Other): Open label study of changes to cellular responses following immunotherapy
  Interventions: Biological: Allergovit grass or birch

INTERVENTIONS:
Biological: Allergovit grass or birch — subcutaneous injection of immunotherapy once weekly for 7 weeks prior to birch pollen season.

SUMMARY:
Hay fever (seasonal allergic rhinitis) results from allergy to grass and tree pollen. The majority of affected individuals manage well with medication from the Pharmacy or from their general practitioner (GP), but for some severely affected people it severely impacts on quality of life. Less than 40% of those affected in UK general practice feel that these medications achieve good symptomatic control.

Specific immunotherapy or desensitisation is the practice of administering small amounts of allergen to allergic patients in increasing doses. This treatment is highly effective in these patients and furthermore is truly disease-modifying, with benefits persisting long-term, even when the treatment has been completed. Desensitisation is a routine treatment in the UK, Europe and North America. The exact immune mechanisms that underlie this symptomatic improvement are not entirely clear. Dr Tarzi, Professor Frew and Professor Kern have recently developed new methods for the investigation of immune responses to allergens. These methods require relatively small blood samples and may provide useful information about how immunotherapy exerts its effects. In addition to improving the investigators basic understanding of this treatment, such knowledge may drive improvements in the treatment and could be useful for monitoring patients for response. The investigators study proposes to investigate changes in the immune responses to pollen allergens during immunotherapy. Blood will be taken just prior to the first immunotherapy injection and again just prior to the final injection. In this way the investigators will be able to compare the immune responses to pollen allergen before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 with no upper age limit
* History of seasonal rhino-conjunctivitis in the appropriate season, not controlled by optimised standard medical therapy
* Positive skin prick test to grass pollen or tree pollen

Exclusion Criteria:

* Inadequately controlled or moderate to severe asthma (GINA III/IV), i.e. the FEV1 is below 70 % of the target value despite adequate pharmacotherapy
* Irreversible changes in the reaction organ (emphysema, bronchiectasis, etc.)
* Clinically significant cardiovascular insufficiency (in cardiovascular diseases, there is an elevated risk of adverse reactions to adrenaline)
* Local or systemic use of beta blockers
* Diseases of the immune system (autoimmune diseases, immune complex-induced immunopathies, immunodeficiencies etc.)
* Malignant disease within the past five years (Patients with previous malignant disease that is considered cured may be included subject to the consent of their oncologist)
* Inability to attend regularly for injections and follow-up visits
* Severe atopic dermatitis
* Pregnant or not using adequate contraception (post-menopausal, surgically sterilised, long-term abstinent, or barrier methods plus spermicide)
* Breast-feeding
* Evidence of current drug or alcohol misuse
* Hypersensitivity to any of the SIT (immunotherapy product) excipients
* Active tuberculosis
* Severe mental disorders
* Multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
What are the changes in T cells associated with immunotherapy? | 6 months
  How does the T cell response change after immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Sussex County Hospital, Brighton, United Kingdom